CLINICAL TRIAL: NCT00608400
Title: Does Dietary Cis-9, Trans-11 Conjugated Linoleic Acid Reduce Parathyroid Hormone in Men?
Brief Title: Effect of Dietary Conjugated Linoleic Acid (CLA) on Parathyroid Hormone in Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Hope Weiler, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HW-08-02; McGill University
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: CLA; PTH; nutritional supplement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): CLA 1.5 g/d
  Interventions: Dietary Supplement: Clarinol CLA
- 2 (Experimental): CLA 3.0 g/d
  Interventions: Dietary Supplement: Clarinol CLA
- 3 (Placebo Comparator)
  Interventions: Dietary Supplement: Clarinol CLA

INTERVENTIONS:
Dietary Supplement: Clarinol CLA — 0, 1.5 or 3.0 g/d dietary conjugated linoleic acids glycerides for 4 months, capsule form

SUMMARY:
The parathyroid gland and its hormone have a major impact on the endocrine control of bone metabolism and mineralization and parathyroid hormone (PTH) has been identified in some epidemiological reports to relate adversely to mortality. Previously, the applicant has demonstrated in two models that dietary cis-9, trans-11 conjugated linoleic acid (CLA) reduces PTH by over 30% in as little as 4 weeks in male rats without adversely affecting bone density. Both bioactive PTH and intact PTH assays have been used and both are reduced by CLA. In one rat model, rats had normal PTH and a sub-group had high PTH due to chronic renal disease. In the second study, the rats were healthy young males and females. Regardless of the model and health state, PTH was reduced 30 to 40% by CLA. Of interest, other isoforms of CLA such as trans-10, cis-12 CLA do not alone result in reduced PTH. The selected CLA isomer proven to reduce PTH, cis-9, trans 11 CLA, is common to food products such as milk fat and beef and is thus more physiologically relevant to the human diet. The global objective of this study is to, for the first time; assess the effects of CLA on PTH in humans, specifically men.

Healthy men 19-53 years of age are selected since bone mass will have reached a peak by this age. Beginning with healthy relatively young men is important versus aging or ill individuals since the effect of CLA on PTH has not been examined and aging and illness might confound the results.

Subjects will be recruited using posters and local newspaper advertisements from the general population. Men (n=30/group) with healthy weights will be randomized to receive 0, 1.5 or 3 g CLA/d for a period of 4 months. At baseline, body weight will be assessed along with whole body bone, lean and fat mass using dual energy x-ray absorptiometry (DXA). Regional bone mass (lumbar spine, total hip, femoral neck) will also be examined using DXA. A blood sample will be taken in the fasted state between 9:00 and 10:00 to examine PTH, ionized Ca, and biomarkers of bone metabolism. After each 1 month on the study, the measurements will be repeated until end of study.

Dietary intake will be monitored along with a survey for possible mild side-effects such as gastrointestinal discomfort. Data will be examined using a mixed model for random (age, weight, vitamin D status) and fixed effects (diet, time) with post-hoc comparisons using Bonferroni correction.

DETAILED DESCRIPTION:
EXPERIMENTAL DETAILS The global objective of this study is to, for the first time; assess the effects of CLA on PTH in humans, specifically men.

Primary Objectives and Hypotheses, in healthy men 40 years of age are to determine if:

1. Cis-9, trans-11 CLA reduces PTH;

   a. it is hypothesized that CLA will reduce PTH by 30%.
2. The effect is transient; b. it is hypothesized that PTH will fall within 4 weeks of treatment and remain stable thereafter over the 4 months of study.
3. Short-term changes in bone metabolism accompany reductions in PTH following dietary intake of CLA; c. it is hypothesized that bone resorption will be reduced as indicated by resorption markers and the ratio of osteoprotegerin to RANKL.

Secondary Objective and Hypothesis is to determine if:

1) Dietary CLA and plasma CLA at baseline are related to bone mass and metabolism;

a. it is hypothesized that higher dietary intakes of CLA and higher plasma CLA will be associated with higher bone mineral density (BMD) and lower bone resorption.

Experimental Design and Methods Population: Healthy men 19 to 53 years of age are selected since bone mass will have reached a peak by this age. Beginning with healthy relatively young men parallels the observations from the animal studies in male rats that were at an age when peak bone mass was already achieved (5 mo). These participants will be recruited from the Greater Montreal area; primarily the Macdonald Campus of McGill University and also through announcements made in the local newspapers (West Island Gazette). All study visits will take place at the Mary Emily Clinical Nutrition Research Unit, School of Dietetics and Nutrition (Directed by Dr. Weiler).

The sample size will be 90 healthy men (n=30/group) based on the following inclusion criteria:

healthy body weight based on body mass index (18.5 - 25 kg/m2 as per Health Canada (50)), no chronic diseases, normal bone mass for age (ie Z-score better than -1 where reference data available), and vitamin D status within optimal range based on serum 25(OH)D (between 50 and 80 nmol/L of serum 25(OH)D with a median threshold of 75 nmol/L as set by international experts (24)).

Vitamin D status will be an inclusion criterion since seasonal changes in vitamin D status will alter PTH. Participants who meet the entry criteria upon screening must also continue to meet the entry criteria 1 month later when the supplementation begins (see figure 3 for flow diagram of study time-line for year 1). This is important as related to vitamin D status and possible interactions with PTH. The error of the vitamin D assay is <10%. Thus measurements at baseline within 10% of the screening value will enable continuance in the study. To ensure that the median threshold is maintained, screening will be set at 75 nmol/L of 25(OH)D and values >10 nmol/L will be accepted at inception. This will accommodate the range set for optimal vitamin D status and is thus 65 nmol/L and up in the present study.

Protocol: In May and June of 2008 potential participants will be initially screened by telephone for health status, self-reported body weight and height and age. Upon meeting these criteria they will be asked to fast beginning the evening prior to the screening visit (12 h) that will include measurement of body weight, height and bone mass using dual-energy x-ray absorptiometry (DXA) to provide whole body and regional bone mass (lumbar spine, total hip, femoral neck) and a general health assessment by the study physicians. At this visit a 5 ml blood sample will be taken between 9 and 10 am to screen for 25(OH)D concentration. It is anticipated that in May-June the 25(OH)D will be within the targeted range in 50-75% of people screened based on the data of Looker et al for US men in northern latitudes in summer where mean values were 79 nmol/L in the northern attitude group of men 40 to 49 years of age (51). Those meeting criteria will be invited to participate in the trial for which men will be randomized to receive 0, 1.5 or 3 g CLA/d for a period of 4 months beginning in ~June of each year; half of the sample will be recruited each year to enable the monthly assessments accompanied by rapid measurement of CLA. Dietary assessment using a 24-hour food recall will establish typical intakes of CLA prior to baseline sampling by mailing the record a week in advance, followed by supplementation. At baseline, body weight and height will be measured along with DXA assessment of whole body and regional bone mass (lumbar spine, forearm, total hip, femoral neck). A food frequency questionnaire will be given to assess the relationship between CLA in the diet, CLA status and bone descriptively. A blood sample will be taken in the fasted state between 9:00 and 10:00 to examine PTH, ionized Ca, and markers of bone metabolism including osteocalcin (formation), osteoprotegerin, RANKL and N-telopeptide (resorption) and CLA in plasma and red cell membranes. This sampling time will accommodate the nadir in PTH as well as permit assessment of biomarkers of bone metabolism at a standardized am time. The measurements (except for the DXA) will be repeated monthly until end of study. Dietary intake will be monitored each month using a 24-hour food recall prior to each visit to enable clarifications in person. A survey for mild side-effects such as gastrointestinal discomfort will be conducted at each visit along with collection of all supplements not taken to estimate compliance. Since participants will be fasting for each visit, a small snack will be provided as tetra pack milk and a bagel after the measurements (under general supplies in budget). Participants will be asked to not exercise prior to the visit since moderately intense activity can elevate PTH (52).

Details of Methodology Dietary Supplementation Approach: All supplements and placebo will be double-blinded by use of letter coding. Only the safety officer will know the treatment groups. Each participant will take the required number of placebo and/or CLA capsules with each lunch and dinner meal and be provided enough for one month at a time. At each visit all unused capsules will be recovered for compliance assessment and a new supply provided for the next month of study. Participants will be asked to maintain their current diet to prevent changes in body weight and body composition and also will be asked to keep their activity as constant as possible over the duration of study, also to keep body weight and composition constant as well as maintain weight bearing activities on bone. Diet will not be modified in this study, but rather monitored. At the screening assessment, a registered dietitian (3 RDs in Dr. Weiler's training program are available to provide this assessment) will provide all participants an assessment of current and usual intake against recommendations and then guide them on how to keep the diet both within recommendations and usual intakes. Participants will be instructed on what amounts of and types of snack foods will be permitted the evening prior to fasting. Of note, calcium intake in Montreal men is typically close to recommendations with ~80% achieving calcium intake at the recommended level (53, 54).

The supplements will be Clarinol A95 (Lipid Nutrition) that is in free fatty acid form with 80% of the CLA in the cis-9, trans-11 form and 20% in the trans-10, cis-12 isoform; this is the purest CLA available. Using supplements for this study is rationalized in order to follow the approach from the basic studies rather than food products enriched with CLA; ie, use diets with the supplemental CLA as used in the rodent study. Each supplement will be designed to provide half of the CLA dosage per meal. In this manner the 1.5 group will have capsules containing 0.75 g of CLA with the remaining weight comprised of placebo olive oil. For the 3 g group, the CLA capsules will contain 1.5 g CLA. The placebo capsules will be olive oil. Each person will be asked to take one half-dose at lunch and one half-dose at dinner.

Dietary and Supplement Intake: will be assessed at each visit using a 24-hour food recall. The data will be used to describe the intakes of the population with respect to total energy, macronutrients (protein, fat, carbohydrate) and micronutrients (Ca, P, Zn, Mg, vitamin D) that relate to bone and PTH metabolism. The food intake for the day prior to blood sampling is also important to establish the possible effects of an evening meal or snack prior to fasting for the am blood sampling. For example if the snack was high in calcium or if the participant did not eat the usual intake etc. values for PTH could be falsely low. The three-day record is selected to better assess intakes and is validated against plasma samples measured for CLA (5, 56). The dietary intake will have less of an impact on the plasma CLA after inception but the dietary intake of CLA is a necessary assessment to demonstrate sources of dietary CLA and to quantify total dietary CLA and enhance understanding of the plasma CLA values.

Sample Procurement: Blood will be collected at all visits between 9:00 and 10:00 to control for diurnal variation permitting 3 to 4 participants to be seen in our Unit daily.

Adverse Effects and Safety Monitoring: At each visit, participants will be asked using a check-box questionnaire if they experienced any illness or been treated for acute illnesses. Frequency of headaches, dizziness, constipation, cramping, nausea, vomiting, diarrhoea or abdominal pain will be documented. Any abnormal value will initiate a second sampling. Upon confirmation of abnormal values, the participant will be asked to stop taking the CLA supplement and have a subsequent blood sample taken at a follow-up visit to evaluate return of ionized Ca and PTH to expected values and they will fall into the intent-to-treat statistical analysis arm of the study. Blood pressure will be measured using standard radial cuff and sphygmomanometer and in supine position immediately following the DXA as part of the general health assessment.

ELIGIBILITY:
Inclusion Criteria:

The sample size will be 90 healthy men (n=30/group) based on the following inclusion criteria:

* Healthy body weight based on body mass index (18.5 - 25 kg/m2 as per Health Canada
* No chronic diseases
* Normal bone mass for age (ie Z-score better than -1 where reference data available)
* Vitamin D status within optimal range based on serum 25(OH)D (between 50 and 80 nmol/L of serum 25(OH)D with a median threshold of 75 nmol/L as set by international experts.

Ages: 19 Years to 53 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Parathyroid Hormone | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Hope A Weiler, PhD, Principal Investigator — McGill University
Locations (1):
- Mary Emily Clinical Nutrition Research Unit, Sainte-Anne-de-Bellevue, Quebec, Canada